CLINICAL TRIAL: NCT05878275
Title: Supporting Infant Development: The Impact of a Tummy Time Intervention on Infant Development
Brief Title: Supporting Infant Development Through Tummy Time, Positioning, and Limiting Baby Gear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-09209-XP
Record Dates: First submitted 2023-03-22; First posted 2023-05-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Prone Position; Child Development
Keywords: Prone Position; Tummy Time; Infant Development

STUDY DESIGN:
Intervention Model Description: Longitudinal experimental design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group Receiving an Informational Tummy Time Brochure (No Intervention): Usual care group will receive a brochure on the importance of tummy time and limiting baby gear.
- Parent Informational Session (Experimental): Parental education session that includes information and a video on avoiding screen time in the first two years of life, the importance and benefits of infants being exposed to tummy time, varying play positions and limiting time in baby gear. Additional information will be provided on the importance of implementing tummy time during the first month of life as well as different ways to implement tummy time and how to increase infant tolerance to tummy time. Parents in the Parent Informational Session can request a Zoom consultation with the Principal Investigator if the parents have questions or need guidance with implementing tummy time.
  Interventions: Behavioral: Parent Informational Session

INTERVENTIONS:
Behavioral: Parent Informational Session — Parents will receive a brochure on the importance of tummy time and limiting baby gear and watch a video on the importance of tummy time and limiting baby gear and receive support for implementing tummy time if requested.
  Arms: Parent Informational Session

SUMMARY:
The goal of this clinical trial is to examine the impact of an educational intervention on infant motor skill development. The main question it aims to answer is: Question 1) Does exposure to an educational intervention on infant development positively impact infant motor skill development? Researchers will compare the intervention group to the treatment as usual group see if there are differences in infant motor skill development.

The purpose of the proposed study is to determine if tummy time, play positions, screen time, and use of baby gear impacts early motor skill development in children. This is a Pilot study. A Pilot study is a small study that is carried out to collect information that will help in the planning of a larger study with the same topic.

DETAILED DESCRIPTION:
The purpose of the proposed study is to examine the impact of an educational intervention on infant motor skill development. A variety of factors influence infant development, including the home environment, maternal education, child rearing practices, caregiver handling, sleep position, baby gear use, and positioning during play. In recent years there have been changes in how babies are positioned when awake. For example, after the American Academy of Pediatrics (AAP) supine sleep recommendation in 1992, some parents reported not placing their infants on the stomach for play (tummy time) while awake due to a fear of sudden infant death syndrome (SIDS). Research suggests that babies who are not exposed to enough tummy time are at risk for delays in the development of their motor skills.

Devices for infant positioning such as swings, bouncy seats, and carriers have also grown in popularity in recent years. More time in containers limits infant mobility and opportunities for exploration and less time in other positions for play. Many parents are not aware that varying how they handle and position their babies can positively influence development, while others have misconceptions about positioning and baby gear use.

Additional research is needed that examines the impact of avoiding screen time, limiting the use of baby gear, regularly implementing tummy time, and varying an infant's position during play. It is also important that parents are aware of the need to initiate tummy time in the first days of life to increase infant tolerance of the position. The following items will constitute as 'baby gear' and will be utilized to determine if their use impacts early motor skill development in children: infant carrier, swing, bouncy seat, or a stationary activity center. The purpose of the proposed study is to determine if an educational intervention on tummy time, play positions, screen time, and use of baby gear impacts early motor skill development in children.

ELIGIBILITY:
Inclusion Criteria:

1. Parent of the infant speaks and reads English
2. Individual is the parent or legal guardian of the infant.
3. Infant is 1 month of age or younger
4. Infant was carried to at least 37-weeks' gestation
5. Parent must own a cell phone will internet access and Zoom or Face Time capability
6. Parent must have a working email address.
7. Parent is over the age of 18 years
8. Family resides within a 30-min driving distance from the University of Tennessee Health Science Center,
9. Infant birthweight of at least 2500 g/ 5.5 pounds
10. Parental report of no know medical condition, health complication or problem since birth
11. that could have an impact on infant movement behaviors or development.
12. Parent reports that infant does not have a diagnosis of Gastroesophageal reflux disease (GERD).
13. Family does not expect to move from the area within 3 years of enrollment

Exclusion Criteria:

1. Infant is regularly cared for by an adult other than their parent for 20 hours or more per week.

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in motor scale score on the Bailey Scales of Infant & Toddler Development | 6 months to 48 months of age
  Scores range from 40 to 160, with higher scores indicating more advanced development

SECONDARY OUTCOMES:
Change in fine motor scale score on the Ages & Stages Questionnaire-3 | 6 months to 48 months of age
  Scores range from 0 to 60 with higher scores indicating more advanced motor development

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Zachry, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are working on a plan to make individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting data will be available upon the acceptance of the research paper. The data will be available for 6 years.
Access Criteria: "Access to data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Result] De Bock F, Braun V, Renz-Polster H. Deformational plagiocephaly in normal infants: a systematic review of causes and hypotheses. Arch Dis Child. 2017 Jun;102(6):535-542. doi: 10.1136/archdischild-2016-312018. Epub 2017 Jan 19. PMID 28104626
- [Result] Dudek-Shriber L, Zelazny S. The effects of prone positioning on the quality and acquisition of developmental milestones in four-month-old infants. Pediatr Phys Ther. 2007 Spring;19(1):48-55. doi: 10.1097/01.pep.0000234963.72945.b1. PMID 17304097
- [Result] Felzer-Kim IT, Erickson K, Adkins C, Hauck JL. Wakeful Prone "Tummy Time" During Infancy: How Can We Help Parents? Phys Occup Ther Pediatr. 2020;40(6):651-668. doi: 10.1080/01942638.2020.1742847. Epub 2020 Mar 19. PMID 32192403
- [Result] Hewitt L, Kerr E, Stanley RM, Okely AD. Tummy Time and Infant Health Outcomes: A Systematic Review. Pediatrics. 2020 Jun;145(6):e20192168. doi: 10.1542/peds.2019-2168. Epub 2020 May 5. PMID 32371428
- [Result] Mendres-Smith AE, Borrero JC, Castillo MI, Davis BJ, Becraft JL, Hussey-Gardner B. Tummy time without the tears: The impact of parent positioning and play. J Appl Behav Anal. 2020 Sep;53(4):2090-2107. doi: 10.1002/jaba.715. Epub 2020 May 20. PMID 32436294
- [Result] Wen LM, Baur LA, Simpson JM, Rissel C, Flood VM. Effectiveness of an early intervention on infant feeding practices and "tummy time": a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Aug;165(8):701-7. doi: 10.1001/archpediatrics.2011.115. PMID 21810633
- [Result] Zachry AH, Kitzmann KM. Caregiver awareness of prone play recommendations. Am J Occup Ther. 2011 Jan-Feb;65(1):101-5. doi: 10.5014/ajot.2011.09100. PMID 21309377
- [Result] Zachry AH, Nolan VG, Hand SB, Klemm SA. Infant Positioning, Baby Gear Use, and Cranial Asymmetry. Matern Child Health J. 2017 Dec;21(12):2229-2236. doi: 10.1007/s10995-017-2344-6. PMID 28725930